CLINICAL TRIAL: NCT01816750
Title: Pilot Study to Assess the Feasibility and Diagnostic Performance of Computed Tomographic Coronary Angiography Using Cardiac Gemstone Spectral Imaging (Cardiac GSI) in Patients With High-risk of Significant Coronary Artery Disease and Myocardial Scar
Brief Title: Cardiac GSI Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 13/P/031; 13/SW/0065 (Other: NRES (UK))
Record Dates: First submitted 2013-02-28; First posted 2013-03-22 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: High Risk of Significant Coronary Artery Disease
Keywords: CT coronary angiography; Coronary disease; Gemstone Spectral Imaging; Diagnostic value; Adaptive statistical iterative reconstruction; iterative reconstruction; Feasibility of coronary and myocardial assessment; novel Cardiac CT GSI protocol
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Anatomical accuracy Cardiac GSI vs ICA (Experimental): The identification and quantification of coronary artery stenoses using Cardiac in comparison to ICA.
  Interventions: Device: Cardiac GSI
- Stress perfusion Cardiac GSI vs MPI-SPECT (Experimental): Assessment of the functional impact of coronary stenoses using Cardiac GSI in comparison to MPI-SPECT
  Interventions: Device: Cardiac GSI
- Delayed enhancement Cardiac GSI vs CMR (Experimental): Assessment of abnormal myocardial tissue characteristics representing ischaemic or scarred tissue using Cardiac GSI in comparison to CMR.
  Interventions: Device: Cardiac GSI

INTERVENTIONS:
Device: Cardiac GSI — A novel method of computed tomography scanning (Cardiac Gemstone Spectral Imaging - Cardiac GSI) and image reconstruction (Adaptive Statistical Iterative Reconstruction- ASIR.
  Other Names: Cardiac Gemstone Spectral Imaging

SUMMARY:
The recently introduced Computed tomography (CT) scanner, Discovery CT750 HD (GE Healthcare, Milwaukee), incorporates a battery of innovations aimed at improving diagnostic image quality, evaluating perfusion and assessing for scar, in an effort to address the current shortcomings of Computed tomographic coronary angiography (CTCA) in patients with significant coronary artery disease. The new scanner will use a novel method of scanning (Cardiac Gemstone Spectral Imaging - Cardiac GSI) and image reconstruction (Adaptive Statistical Iterative Reconstruction- ASIR) as opposed to standard definition 64-slice CT Multi-detector row computed tomography(MDCT)and Filtered Back Projection (FBP) used by the conventional CT scanners. The Cardiac GSI protocol enables the scanner to acquire images at two different x-ray energies almost simultaneously, which can be post-processed to selectively reduce beam hardening artefacts and delete materials with specific attenuating properties from the images, such as coronary calcium. ASIR offsets the potential increase in radiation dose required for Cardiac GSI scanning. This will potentially result in images of higher diagnostic quality with an equivalent or perhaps lower dose of radiation compared to present technology.

Furthermore, it is hypothesised that dual-energy acquisition may improve the accuracy of the assessment of perfusion.

Although initial in-vitro results are encouraging, this technology has not been rigorously assessed with regards to its feasibility and diagnostic quality, limiting its applicability in routine clinical practice. This assessment will require a trial comparing the accuracy of Cardiac GSI CTCA with that of Invasive coronary angiography (ICA) for anatomical assessment of stenosis, Myocardial Perfusion Imaging with Single Photon Emission Computed Tomography (MPI-SPECT) for assessment of perfusion and Cardiac Magnetic Resonance (CMR) for assessment of myocardial scar. We have designed a pilot study in this regard which will help us assess the feasibility of the scan protocol and provide data to power a larger study to assess the diagnostic remit of Cardiac GSI scanning in the assessment of patients with high-risk of significant coronary artery disease and myocardial scar.

ELIGIBILITY:
Inclusion Criteria:

Accuracy arm

* Patients >50 years of age
* Suspected or known coronary artery disease referred for ICA

Stress perfusion arm

* Patients >50 years of age
* Suspected or established coronary artery disease referred for MPI-SPECT for assessment of inducible ischaemia

Delayed enhancement arm

* Patients >50 years of age
* Referred for CMR for assessment of myocardial viability/scar

Exclusion Criteria:

Accuracy arm

* Consent cannot be obtained
* Patient BMI > 30 kg /m2
* NYHA class III or IV heart failure
* Chronic total occlusion of target epicardial coronary artery
* Urgent revascularisation required
* Allergy to iodinated contrast or previous contrast induced nephropathy
* Intolerance or contraindication to beta-blockers
* Uncontrolled heart rhythm disturbances
* 2nd or 3rd degree atrioventricular block
* Estimated glomerular filtration rate <30ml/min within two weeks prior to procedure or chronic renal failure on dialysis
* Pregnancy

Stress perfusion arm

* As above, plus:
* Asthma (any) or intolerance to adenosine

Delayed enhancement arm

- As for Accuracy arm

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Feasibility - Assessment of rates of recruitment, acceptability of the procedure to patients, ease of CT acquisition | 4 months
  Assessment of rates of recruitment, acceptability of the procedure to patients, ease of CT acquisition. This pilot study will add to this assessment with specific information about the diagnostic performance of the novel scanning technique:
  * Are images of sufficient quality to be diagnostic?
  * Is diagnosis likely to be non-inferior to current comparable techniques, sufficient to justify a formal study?

SECONDARY OUTCOMES:
radiation burden of the Cardiac GSI techniques | 4 months
  The Discovery CT750 HD scanner uses a new image reconstruction technique called Adaptive Statistical Iterative Reconstruction (ASIR). ASIR uses more complex mathematical modelling for image reconstruction, thus reducing the need for statistical assumptions and reducing image noise and artefact. It also requires the less raw data and thus significantly less radiation dose. Studies suggest that using ASIR can achieve up to 40% dose reduction compared to Filtered Back Projection (FBP).
  However, the effect of ASIR and radiation dose reducing algorithms on image quality and accuracy has not been assessed and the difference in image quality and artefact suppression using the new technology remains to be established before its widespread dissemination into clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Clayton, MBBS, Principal Investigator — Plymouth Hospitals NHS Trust (UK); Gareth Morgan-Hughes, MBBS, Principal Investigator — Plymouth Hospitals NHS Trust (UK); Franchesca Wotton, MBBS, Study Director — Plymouth Hospitals NHS Trust (UK)
Locations (1):
- Plymouth Hospitals NHS Trust, Plymouth, Devon, United Kingdom